CLINICAL TRIAL: NCT06279117
Title: The Effect of Therapeutic Touch Applied to Nursing Students on Exam Anxiety
Brief Title: The Effect of Therapeutic Touch on Exam Anxiety
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dokuz Eylul University (Other)
Responsible Party: Principal Investigator, Gizem Göktuna, Principal Investigator, Dokuz Eylul University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2023/9/8
Record Dates: First submitted 2024-02-18; First posted 2024-02-26 (Actual); Last update posted 2024-05-21 (Actual); Status verified 2024-05

CONDITIONS: Test Anxiety
Keywords: therapeutic touch; nursing care; test anxiety
MeSH Terms: interventions — Therapeutic Touch

STUDY DESIGN:
Intervention Model Description: Randomised controlled clinical trial
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Therapeutic touch group (Experimental): Individuals who undergo therapeutic touch will receive therapeutic touch for 20 minutes 30 minutes before the exam.
  Interventions: Behavioral: therapeutic touch
- control group (No Intervention): No treatment will be performed on individuals in the control group.

INTERVENTIONS:
Behavioral: therapeutic touch — Individuals who undergo therapeutic touch will receive therapeutic touch for 20 minutes 30 minutes before the exam.
  Arms: Therapeutic touch group

SUMMARY:
Aim: This study was planned to determine the effect of therapeutic touch applied to nursing students on test anxiety.

Method: Students who met the inclusion criteria were divided into therapeutic touch and control groups using the randomization method. After the groups were determined, the students filled out the Introductory Information Form and the State Exam Anxiety Scale. 30 minutes before the exam, therapeutic touch was applied to each of the students, who were divided into groups, for 20 minutes. No application was made to the control group, and they were told to wait in the classroom where the group was waiting as they wished.Immediately after the application was completed, the scale was re-applied to both groups.

DETAILED DESCRIPTION:
Test anxiety is a condition that has cognitive, emotional and physiological aspects and causes unwanted and disturbing emotions during the exam. It can inhibit the mental perception needed to do well on an exam, as well as the clear thinking skills and memory needed to study effectively.The person may feel anxious, worthless or disorganized, experience rapid heartbeat, headaches and stress; They may compare themselves with their peers due to test anxiety. Test anxiety can hinder educational success and negatively impact students' skill development and academic performance. Nursing education is a highly stressful process that includes theoretical and practical learning and teaching experiences. This situation further increases students' anxiety levels. Studies have found that nursing students' test anxiety is higher than other university students.I t is known that many complementary methods are used to reduce anxiety. Therapeutic touch, which is one of the energy-based practices, is one of them.

When the literature is examined, it can be seen that therapeutic touch has been studied on symptoms such as anxiety, fatigue, sleep quality, comfort and pain in different sample groups, but there is no study on test anxiety.Therefore, this study was planned to determine the effect of therapeutic touch applied to nursing students on test anxiety.

ELIGIBILITY:
Inclusion Criteria:

* To be over 18 years of age,
* To know Turkish and to agree to participate in the research
* Being a fourth year nursing student
* Not having received any energy therapy (reiki, therapeutic touch) before

Exclusion Criteria:

* Presence of existing psychiatric illness,
* Using anxiolytic and antidepressant medications

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 46 (Actual)
Dates: Start 2024-01-15 (Actual); Primary Completion 2024-05-15 (Actual); Study Completion 2024-05-18 (Actual)

PRIMARY OUTCOMES:
Text Anxiety | Individuals in the therapeutic touch and control groups will be measured as a baseline before the application.
  Comparison of test anxiety results of therapeutic touch group and control group. The students' test anxiety score data were collected by the State Test Anxiety Scale.
  It is a 22-item scale. The scores in the inventory range from 22 to 88. Higher points show a higher level of anxiety.
Text Anxiety | After the therapeutic touch is completed, individuals in both groups will be measured again within an average of 10 minutes.
  Comparison of test anxiety results of therapeutic touch group and control group. The students' test anxiety score data were collected by the State Test Anxiety Scale.
  It is a 22-item scale. The scores in the inventory range from 22 to 88. Higher points show a higher level of anxiety.

CONTACTS AND LOCATIONS:
Locations (1):
- Gizem Göktuna, Izmir, Turkey (Türkiye)